CLINICAL TRIAL: NCT02478996
Title: Internet-based Perioperative Exercise Program in Patients With Barrett's Carcinoma Scheduled for Esophagectomy (iPEP Study) A Prospective Randomized-controlled Pilot Trial
Brief Title: Internet-based Perioperative Exercise Program in Patients With Barrett's Carcinoma Scheduled for Esophagectomy
Acronym: iPEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Dr. Ines Gockel, Prof. Dr., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFSM-01
Record Dates: First submitted 2015-05-26; First posted 2015-06-23 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Barrett Esophagus
Keywords: perioperative; internet-based; exercise program
MeSH Terms: conditions — Barrett Esophagus

ARMS (2):
- Internet-based exercise program (Experimental): The intervention group is supervised by a sports scientist eight to twelve weeks before and after surgery. Patients receive an individually designed intensive exercise program based on the functional and Fitness measurements at first diagnosis.
  Interventions: Other: Internet-based exercise program
- Basis therapy (No Intervention): Participants of the Treatment as usual (TAU) group receive written information material enlightening the importance of regular physical activities and general releases on preparation for esophagectomy.

INTERVENTIONS:
Other: Internet-based exercise program — Patients undergo internet-based perioperative exercise program (iPEP), including daily endurance, resistance and ventilation training
  Arms: Internet-based exercise program

SUMMARY:
This study will evaluate, if an intensive individually adaptated training program via online supervision during neoadjuvant therapy will improve lung function and reduce pulmonary complications following esophagectomy for Barrett's cancer.

DETAILED DESCRIPTION:
Patients undergoing surgery for esophageal cancer have a high risk for postoperative deterioration of lung function and pulmonal complications. This may be partly due to one-lung ventilation during the thoracic part of the operation. This often encounters for prolonged periods of reconvalescence and reduced quality of life, apart from socioeconomic disadvantages. Physical preconditioning has become a crucial leverage to optimize fitness and lung function in patients scheduled for esophagectomy, in particular during the interval of neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the esophagus or adenocarcinoma of the esophagogastric junction type I according to Siewert's classification, clinical stages IIB-IIIC (T3/T4 and/or N+; M0) according to Union Internationale Contre le Cancer (UICC), 7th Edition
* Resectable stage according to discussion in the local multidisciplinary tumor board (MDT) of the participating centers and patient medically fit for multimodality therapy (ECOG performance status at least 1 or better, no severe impairment of cardiac, renal, hepatic, endocrine, bone marrow and cerebral functions)
* Planned abdominal-thoracic esophagectomy with gastric pull-up and intrathoracic or cervical anastomosis
* Cognitive ability of the patient to understand the perioperative program and to participate actively

Exclusion Criteria:

* Presence of a second malignant tumor (unless curatively treated > 5 years ago)
* Chemotherapy or radiochemotherapy in patient's history
* Orthopedic, rheumatologic, cardiovascular or neurologic (epilepsy, stroke, Parkinson's disease, muscle wasting diseases such as amyotrophic lateral sclerosis or multiple sclerosis) contraindications for the sports program
* Inability to use the internet or no internet Access
* Inability to communicate in German
* Each active disease, which hinders completion of the study
* Active alcoholism or illegal drug consumption within the last six months before study entry

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
peak oxygen uptake (VO2peak) | 6 months
  First measurement three months prior to surgery (baseline), Second measurement immediately before surgery, third measurement three months after esophagectomy

SECONDARY OUTCOMES:
Gastric conduit failure after esophagectomy | intraoperative
  (type classification according to Veeramootoo et al. (2009)) Evaluation of postoperative in-hospital stay
pneumonia | intraoperative
  Evaluation of postoperative in-hospital stay
duration of mechanical ventilation | intraoperative
  Evaluation of postoperative in-hospital stay
re-intubation rate | intraoperative
  Evaluation of postoperative in-hospital stay
Duration of intensive care unit stay | intraoperative
  Evaluation of postoperative in-hospital stay
quality of life | 6 months
  Quality of life questionnaire (QoLQ-C30) with the esophagus-specific module OES-18. First measurement three months prior to surgery (baseline), immediately before surgery, three months after esophagectomy

OTHER OUTCOMES:
feasibility of the online-based sports program | 6 months
  analysis by written questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Perikles Simon, Prof.Dr.Dr., Principal Investigator — Department of Sports Medicine, Disease Prevention and Rehabilitation, Johannes Gutenberg-University of Mainz; Ines Gockel, Prof. Dr., Principal Investigator — Department of Visceral, Transplantation, Vascular and Thoracic Surgery, University Hospital of Leipzig
Locations (1):
- Department of Visceral, Transplantation, Vascular and Thoracic Surgery, Leipzig, Germany

REFERENCES:
- [Background] Gockel I, Niebisch S, Ahlbrand CJ, Hoffmann C, Mohler M, Duber C, Lang H, Heid F. Risk and Complication Management in Esophageal Cancer Surgery: A Review of the Literature. Thorac Cardiovasc Surg. 2016 Oct;64(7):596-605. doi: 10.1055/s-0034-1399763. Epub 2015 Jan 28. PMID 25629461
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Derogar M, Orsini N, Sadr-Azodi O, Lagergren P. Influence of major postoperative complications on health-related quality of life among long-term survivors of esophageal cancer surgery. J Clin Oncol. 2012 May 10;30(14):1615-9. doi: 10.1200/JCO.2011.40.3568. Epub 2012 Apr 2. PMID 22473157
- [Background] Biere SS, van Berge Henegouwen MI, Maas KW, Bonavina L, Rosman C, Garcia JR, Gisbertz SS, Klinkenbijl JH, Hollmann MW, de Lange ES, Bonjer HJ, van der Peet DL, Cuesta MA. Minimally invasive versus open oesophagectomy for patients with oesophageal cancer: a multicentre, open-label, randomised controlled trial. Lancet. 2012 May 19;379(9829):1887-92. doi: 10.1016/S0140-6736(12)60516-9. Epub 2012 May 1. PMID 22552194
- [Background] Schwenk W. [Fast track rehabilitation in visceral surgery]. Chirurg. 2009 Aug;80(8):690-701. doi: 10.1007/s00104-009-1676-1. German. PMID 19568723
- [Background] Bardram L, Funch-Jensen P, Jensen P, Crawford ME, Kehlet H. Recovery after laparoscopic colonic surgery with epidural analgesia, and early oral nutrition and mobilisation. Lancet. 1995 Mar 25;345(8952):763-4. doi: 10.1016/s0140-6736(95)90643-6. PMID 7891489
- [Background] Cerfolio RJ, Bryant AS, Bass CS, Alexander JR, Bartolucci AA. Fast tracking after Ivor Lewis esophagogastrectomy. Chest. 2004 Oct;126(4):1187-94. doi: 10.1378/chest.126.4.1187. PMID 15486381
- [Background] Cao S, Zhao G, Cui J, Dong Q, Qi S, Xin Y, Shen B, Guo Q. Fast-track rehabilitation program and conventional care after esophagectomy: a retrospective controlled cohort study. Support Care Cancer. 2013 Mar;21(3):707-14. doi: 10.1007/s00520-012-1570-0. Epub 2012 Aug 30. PMID 22933129
- [Background] Jensen LS, Pilegaard HK, Eliasen M, Mehlsen NC, Kehlet H. [Esophageal resection in an accelerated postoperative recovery regimen]. Ugeskr Laeger. 2004 Jun 21;166(26-31):2560-3. No abstract available. Danish. PMID 15285164
- [Background] Neal JM, Wilcox RT, Allen HW, Low DE. Near-total esophagectomy: the influence of standardized multimodal management and intraoperative fluid restriction. Reg Anesth Pain Med. 2003 Jul-Aug;28(4):328-34. doi: 10.1016/s1098-7339(03)00197-4. PMID 12945027
- [Background] Blom RL, van Heijl M, Bemelman WA, Hollmann MW, Klinkenbijl JH, Busch OR, van Berge Henegouwen MI. Initial experiences of an enhanced recovery protocol in esophageal surgery. World J Surg. 2013 Oct;37(10):2372-8. doi: 10.1007/s00268-013-2135-1. PMID 23807122
- [Background] Veeramootoo D, Parameswaran R, Krishnadas R, Froeschle P, Cooper M, Berrisford RG, Wajed SA. Classification and early recognition of gastric conduit failure after minimally invasive esophagectomy. Surg Endosc. 2009 Sep;23(9):2110-6. doi: 10.1007/s00464-008-0233-1. Epub 2008 Dec 6. PMID 19067058
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Kondrup J, Allison SP, Elia M, Vellas B, Plauth M; Educational and Clinical Practice Committee, European Society of Parenteral and Enteral Nutrition (ESPEN). ESPEN guidelines for nutrition screening 2002. Clin Nutr. 2003 Aug;22(4):415-21. doi: 10.1016/s0261-5614(03)00098-0. PMID 12880610
- [Background] Martin L, Birdsell L, Macdonald N, Reiman T, Clandinin MT, McCargar LJ, Murphy R, Ghosh S, Sawyer MB, Baracos VE. Cancer cachexia in the age of obesity: skeletal muscle depletion is a powerful prognostic factor, independent of body mass index. J Clin Oncol. 2013 Apr 20;31(12):1539-47. doi: 10.1200/JCO.2012.45.2722. Epub 2013 Mar 25. PMID 23530101
- [Background] Trappe HJ, Lollgen H. [Guidelines for ergometry. German Society of Cardiology--Heart and Cardiovascular Research]. Z Kardiol. 2000 Sep;89(9):821-31. doi: 10.1007/s003920070190. No abstract available. German. PMID 11077695
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Kinugasa S, Tachibana M, Yoshimura H, Ueda S, Fujii T, Dhar DK, Nakamoto T, Nagasue N. Postoperative pulmonary complications are associated with worse short- and long-term outcomes after extended esophagectomy. J Surg Oncol. 2004 Nov 1;88(2):71-7. doi: 10.1002/jso.20137. PMID 15499604
- [Background] Kumagai K, Rouvelas I, Tsai JA, Mariosa D, Klevebro F, Lindblad M, Ye W, Lundell L, Nilsson M. Meta-analysis of postoperative morbidity and perioperative mortality in patients receiving neoadjuvant chemotherapy or chemoradiotherapy for resectable oesophageal and gastro-oesophageal junctional cancers. Br J Surg. 2014 Mar;101(4):321-38. doi: 10.1002/bjs.9418. Epub 2014 Feb 3. PMID 24493117
- [Background] Rock CL, Doyle C, Demark-Wahnefried W, Meyerhardt J, Courneya KS, Schwartz AL, Bandera EV, Hamilton KK, Grant B, McCullough M, Byers T, Gansler T. Nutrition and physical activity guidelines for cancer survivors. CA Cancer J Clin. 2012 Jul-Aug;62(4):243-74. doi: 10.3322/caac.21142. Epub 2012 Apr 26. PMID 22539238
- [Background] Fletcher GF, Balady GJ, Amsterdam EA, Chaitman B, Eckel R, Fleg J, Froelicher VF, Leon AS, Pina IL, Rodney R, Simons-Morton DA, Williams MA, Bazzarre T. Exercise standards for testing and training: a statement for healthcare professionals from the American Heart Association. Circulation. 2001 Oct 2;104(14):1694-740. doi: 10.1161/hc3901.095960. No abstract available. PMID 11581152
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Watson YI, Arfken CL, Birge SJ. Clock completion: an objective screening test for dementia. J Am Geriatr Soc. 1993 Nov;41(11):1235-40. doi: 10.1111/j.1532-5415.1993.tb07308.x. PMID 8227899
- [Result] Valkenet K, van de Port IG, Dronkers JJ, de Vries WR, Lindeman E, Backx FJ. The effects of preoperative exercise therapy on postoperative outcome: a systematic review. Clin Rehabil. 2011 Feb;25(2):99-111. doi: 10.1177/0269215510380830. Epub 2010 Nov 8. PMID 21059667
- [Result] Feeney C, Reynolds JV, Hussey J. Preoperative physical activity levels and postoperative pulmonary complications post-esophagectomy. Dis Esophagus. 2011 Sep;24(7):489-94. doi: 10.1111/j.1442-2050.2010.01171.x. Epub 2011 Feb 10. PMID 21309920
- [Result] Tatematsu N, Park M, Tanaka E, Sakai Y, Tsuboyama T. Association between physical activity and postoperative complications after esophagectomy for cancer: a prospective observational study. Asian Pac J Cancer Prev. 2013;14(1):47-51. doi: 10.7314/apjcp.2013.14.1.47. PMID 23534776
- [Result] van Adrichem EJ, Meulenbroek RL, Plukker JT, Groen H, van Weert E. Comparison of two preoperative inspiratory muscle training programs to prevent pulmonary complications in patients undergoing esophagectomy: a randomized controlled pilot study. Ann Surg Oncol. 2014 Jul;21(7):2353-60. doi: 10.1245/s10434-014-3612-y. Epub 2014 Mar 7. PMID 24604584
- [Result] Dettling DS, van der Schaaf M, Blom RL, Nollet F, Busch OR, van Berge Henegouwen MI. Feasibility and effectiveness of pre-operative inspiratory muscle training in patients undergoing oesophagectomy: a pilot study. Physiother Res Int. 2013 Mar;18(1):16-26. doi: 10.1002/pri.1524. Epub 2012 Apr 10. PMID 22489016
- [Result] Agrelli TF, de Carvalho Ramos M, Guglielminetti R, Silva AA, Crema E. Preoperative ambulatory inspiratory muscle training in patients undergoing esophagectomy. A pilot study. Int Surg. 2012 Jul-Sep;97(3):198-202. doi: 10.9738/CC136.1. PMID 23113846
- [Result] Inoue J, Ono R, Makiura D, Kashiwa-Motoyama M, Miura Y, Usami M, Nakamura T, Imanishi T, Kuroda D. Prevention of postoperative pulmonary complications through intensive preoperative respiratory rehabilitation in patients with esophageal cancer. Dis Esophagus. 2013 Jan;26(1):68-74. doi: 10.1111/j.1442-2050.2012.01336.x. Epub 2012 Mar 12. PMID 22409435
- [Result] Valkenet K, Trappenburg JC, Gosselink R, Sosef MN, Willms J, Rosman C, Pieters H, Scheepers JJ, de Heus SC, Reynolds JV, Guinan E, Ruurda JP, Rodrigo EH, Nafteux P, Fontaine M, Kouwenhoven EA, Kerkemeyer M, van der Peet DL, Hania SW, van Hillegersberg R, Backx FJ. Preoperative inspiratory muscle training to prevent postoperative pulmonary complications in patients undergoing esophageal resection (PREPARE study): study protocol for a randomized controlled trial. Trials. 2014 Apr 27;15:144. doi: 10.1186/1745-6215-15-144. PMID 24767575
- [Derived] Pfirrmann D, Haller N, Huber Y, Jung P, Lieb K, Gockel I, Poplawska K, Schattenberg JM, Simon P. Applicability of a Web-Based, Individualized Exercise Intervention in Patients With Liver Disease, Cystic Fibrosis, Esophageal Cancer, and Psychiatric Disorders: Process Evaluation of 4 Ongoing Clinical Trials. JMIR Res Protoc. 2018 May 22;7(5):e106. doi: 10.2196/resprot.8607. PMID 29789277
- [Derived] Pfirrmann D, Tug S, Brosteanu O, Mehdorn M, Busse M, Grimminger PP, Lordick F, Glatz T, Hoeppner J, Lang H, Simon P, Gockel I. Internet-based perioperative exercise program in patients with Barrett's carcinoma scheduled for esophagectomy [iPEP - study] a prospective randomized-controlled trial. BMC Cancer. 2017 Jun 14;17(1):413. doi: 10.1186/s12885-017-3400-8. PMID 28615010